CLINICAL TRIAL: NCT05470556
Title: Investigation of Peak Expiratory Flow, Physical Activity Level, Anthropometric Measurements, and Core Performance in Obese and Overweight Adolescents
Brief Title: Investigation of Peak Expiratory Flow and Physically Fitness in Obese and Overweight Adolescents
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc. Prof., Biruni University
Other Study IDs: 2022/70-09
Record Dates: First submitted 2022-06-24; First posted 2022-07-22 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
Keywords: peak expiratory flow; core muscle strength; physical activity
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Overweight adolescents: This group will consist of 20 overweight adolescents (Body mass index (BMI) percentile value is 85.-95)
- Obese adolescents: This group will consist of 20 obese adolescents (BMI percentile value is above the 95th)
- normal weight: This group will consist of 20 normal-weight adolescents (BMI percentile value is 5th-85th.)

SUMMARY:
Due to the increasing prevalence of childhood obesity and overweight, health problems may begin to appear at an early age. The aim of this study is to examine physical activity level, core performance, anthropometric measurements and peak expiratory flow in overweight and obese adolescents compared to normal weight adolescents.

DETAILED DESCRIPTION:
Due to the increasing prevalence of childhood obesity and overweight, health problems may begin to appear at an early age. Overweight and obese people are at risk for medical conditions that can lead to greater morbidity and mortality. Lack of physical activity is a well-known risk factor for obesity and the relationship between them has been supported by many studies. It has also been reported by studies that obesity affects respiratory parameters. In overweight and obese adolescents, a relationship is likely between the affected respiratory parameters and the weakened core region. There are not enough studies on this subject in the literature. Therefore, the aim of the study is to examine the physical activity level, core performance, anthropometric measurements and peak expiratory flow in overweight and obese adolescents in comparison with normal weight adolescents.

ELIGIBILITY:
* Inclusion Criteria for the Obese and Overweight Group:
* BMI percentile value is 85.-95. between and above the 95th,
* Do not have any chronic disease,
* Do not have orthopedic problems that would prevent them from participating in the study,
* Secondary school students who are willing to participate in the study and whose parents' consent has been obtained will be included.
* Inclusion Criteria for the Normal Weight Group:
* BMI percentile value is 5th-85th. between,
* Do not have any chronic disease,
* Having no orthopedic and neurological problems that would prevent them from participating in the study,
* Secondary school students who are willing to participate in the study and whose parents' consent has been obtained will be included.
* Exclusion Criteria:
* BMI percentile value below the 5th,
* With chronic cardiac and pulmonary disease,
* Having a diagnosis of neurological or other disease affecting cognitive functions,
* Individuals receiving medical treatment that will affect attention and concentration will not be included.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will consist of 60 volunteer adolescents who are obese, overweight and normal weight studying in the 5th, 6th and 7th grades of secondary school.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow (PEF) | baseline
  Peak expiratory flow will be measured with a peak expiratory flow meter. The measurement is taken while the person is standing. After taking a deep breath, exhale as hard and as fast as you can. 3 measurements will be made and the best value will be recorded as peak expiratory flow-PEF (L/min).

SECONDARY OUTCOMES:
Core Muscle Strength | baseline
  A modified push-up and sit-up test will be used to evaluate the strength of the core muscles. Measurements will be made using a stopwatch and the number of repetitions in 30 seconds will be recorded.
Child Physical Activity Questionnaire | baseline
  Only 9 of the 10 items that make up the scale are used to calculate activity scores. Evaluates the activities done for 7 days. It consists of 5 stages of scoring. 1 indicates the lowest, 5 the highest level of physical activity. The average of the total score indicates the summary score. A higher score indicates a higher level of physical activity.
Neck circumference | baseline
  Neck circumference will be measured from the lower border of the laryngeal protrusion with a tape measure.
Waist circumference | baseline
  Waist circumference will be measured with a tape measure in the standing position, by determining the midpoint between the lowest rib and the iliac crest from the exposed waist circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, PT, PhD, Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No